CLINICAL TRIAL: NCT01219244
Title: Enhancing Memory Functions in Patients With Mild Cognitive Impairment by Dietary Interventions and in Combination With Exercise and Cognitive Training - Proof of Concept and Mechanisms
Brief Title: Effects of Dietary Interventions on the Brain in Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr. med. Agnes Flöel, Neurologie, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: nutrition_memory_01
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Mild Cognitive Impairment
Keywords: memory; diet; elderly; cognition; prevention; lifestyle
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Caloric Restriction; Restraint, Physical; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Caloric restriction (Experimental)
  Interventions: Behavioral: caloric restriction
- omega-3 supplementation (Experimental)
  Interventions: Behavioral: omega-3 supplementation
- resveratrol supplementation (Experimental)
  Interventions: Behavioral: resveratrol supplementation
- placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo
- 2nd step: intervention + physical /cognitive training (Experimental): most effective dietary intervention plus physical and cognitive training
  Interventions: Behavioral: 2nd step: intervention + physical / cognitive training
- 2nd step: most effective dietary intervention plus control (Placebo Comparator): most effective dietary intervention plus control
  Interventions: Behavioral: 2nd step: intervention + control

INTERVENTIONS:
Behavioral: caloric restriction — 6 months of caloric restriction (15 %)
  Arms: Caloric restriction
Behavioral: omega-3 supplementation — 6 months of omega-3 supplementation
  Arms: omega-3 supplementation
Behavioral: resveratrol supplementation — 6 months of resveratrol supplementation
  Arms: resveratrol supplementation
Behavioral: Placebo — 6 months of placebo intake
  Arms: placebo
Behavioral: 2nd step: intervention + physical / cognitive training — most effective dietary intervention plus physical and cognitive training
  Arms: 2nd step: intervention + physical /cognitive training
Behavioral: 2nd step: intervention + control — most effective dietary intervention plus control
  Arms: 2nd step: most effective dietary intervention plus control

SUMMARY:
The study will investigate whether dietary modification could provide positive effects on brain functions in elderly people with mild cognitive impairment.

DETAILED DESCRIPTION:
The age-related degradation of cognitive functions even to the point of neurodegenerative disorders such as Alzheimer's disease are a growing public-health concern with devastating effects.

Referring to animal data, empirical studies, and pilot human trials, dietary modification (caloric restriction, omega-3 fatty acids and resveratrol) should improve cognitive functions such as learning and memory. To test this hypothesis, the researchers study general brain functions in elderly subjects (50-80 years old) with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* subjects with mild cognitive impairment
* 50-80 years old
* moderate to heavy weight (BMI 25-35)

Exclusion Criteria:

* dementia
* diabetes
* severe disease
* younger than 50 years
* BMI < 25

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - cognitive subscale | Prior to intervention and after 6 months of intervention

SECONDARY OUTCOMES:
Functional/Structural brain changes | Prior to intervention and after 6 months of intervention
Plasma biomarkers | Prior to intervention and after 6 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof., Study Chair — Charité University Berlin
Locations (1):
- Department of Neurology, Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Kobe T, Witte AV, Schnelle A, Lesemann A, Fabian S, Tesky VA, Pantel J, Floel A. Combined omega-3 fatty acids, aerobic exercise and cognitive stimulation prevents decline in gray matter volume of the frontal, parietal and cingulate cortex in patients with mild cognitive impairment. Neuroimage. 2016 May 1;131:226-38. doi: 10.1016/j.neuroimage.2015.09.050. Epub 2015 Oct 1. PMID 26433119
- [Result] Kobe T, Witte AV, Schnelle A, Tesky VA, Pantel J, Schuchardt JP, Hahn A, Bohlken J, Grittner U, Floel A. Impact of Resveratrol on Glucose Control, Hippocampal Structure and Connectivity, and Memory Performance in Patients with Mild Cognitive Impairment. Front Neurosci. 2017 Mar 7;11:105. doi: 10.3389/fnins.2017.00105. eCollection 2017. PMID 28326010
- [Result] Witte AV, Kobe T, Graunke A, Schuchardt JP, Hahn A, Tesky VA, Pantel J, Floel A. Impact of leptin on memory function and hippocampal structure in mild cognitive impairment. Hum Brain Mapp. 2016 Dec;37(12):4539-4549. doi: 10.1002/hbm.23327. Epub 2016 Aug 11. PMID 27511061
- [Result] Wirth M, Pichet Binette A, Brunecker P, Kobe T, Witte AV, Floel A. Divergent regional patterns of cerebral hypoperfusion and gray matter atrophy in mild cognitive impairment patients. J Cereb Blood Flow Metab. 2017 Mar;37(3):814-824. doi: 10.1177/0271678X16641128. Epub 2016 Jul 20. PMID 27037094
- [Result] Kobe T, Witte AV, Schnelle A, Grittner U, Tesky VA, Pantel J, Schuchardt JP, Hahn A, Bohlken J, Rujescu D, Floel A. Vitamin B-12 concentration, memory performance, and hippocampal structure in patients with mild cognitive impairment. Am J Clin Nutr. 2016 Apr;103(4):1045-54. doi: 10.3945/ajcn.115.116970. Epub 2016 Feb 24. PMID 26912492